CLINICAL TRIAL: NCT04898049
Title: Suicide Risk Within 30 Days After a Potentially Traumatic Event (PTE) in Patients Treated by a Medico-psychological Emergency Unit. Prospective Cohort Study
Brief Title: Suicide Risk 30 Days After a Potentially Traumatic Event in Patients Treated by a Medico-psychological Emergency Unit
Acronym: SCAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.398
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Suicide Risk
Keywords: Suicide risk; potentially traumatic event; medico-psychological emergency unit; 30 days

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The national french survey "Mental health in general population", showed that the risk of suicide was significantly increased during exposure to a potentially traumatic event (PTE), with an increasing gradient depending on the psychological impact. This included not only people suffering from post-traumatic stress disorder but also those confronted with PTE, presenting or having presented phenomena of reviviscence or at least an element of psychopathological impact. This risk could concern 30.2% of the population over the entire lifetime. Internationally, recent reviews of the literature tend to show that victims of interpersonal violence are more at risk of suicide (OR 1.99 95% CI: 1.73-2.28). Nevertheless, the literature remains heterogeneous, the definitions vague and the temporal proximity of the violence little taken into account. It is therefore a large-scale phenomenon that remains little explored.

To increase our knowledge in this area, the investigators will focus on patients treated by Emergency Medical Psychological Cells (CUMP), that is victims of disasters, accidents involving a large number of victims or events that may have significant psychological repercussions due to the circumstances surrounding them.

DETAILED DESCRIPTION:
The national french survey "Mental health in general population", showed that the risk of suicide was significantly increased during exposure to a potentially traumatic event (PTE), with an increasing gradient depending on the psychological impact. This included not only people suffering from post-traumatic stress disorder but also those confronted with PTE, presenting or having presented phenomena of reviviscence or at least an element of psychopathological impact. This risk could concern 30.2% of the population over the entire lifetime. Internationally, recent reviews of the literature tend to show that victims of interpersonal violence are more at risk of suicide (OR 1.99 95% CI: 1.73-2.28). Nevertheless, the literature remains heterogeneous, the definitions vague and the temporal proximity of the violence little taken into account. It is therefore a large-scale phenomenon that remains little explored.

To increase our knowledge in this area, the investigators will focus on patients treated by Emergency Medical Psychological Cells (CUMP), that is victims of disasters, accidents involving a large number of victims or events that may have significant psychological repercussions due to the circumstances surrounding them.

Estimate the prevalence of suicide risk 30 days after exposure to a potentially traumatic event, in people treated by a CUMP

The secondary objective aim to identify:

1. The main psychiatric disorders at 30 days (depressive disorders, bipolar disorders, panic disorder, agoraphobia, social phobia, generalized anxiety, post-traumatic stress disorder, obsessive-compulsive disorder, disorder linked to the consumption of alcohol or other substances, psychotic disorders, eating disorders)
2. The number of death by suicide 1 year after the trauma
3. The incidence of suicide attempts 1 year after the trauma
4. The incidence of suicidal ideation 1 year of trauma Prognostic factors of mortality by suicide, suicide attempts or suicidal ideation will be sought.

A number of 215 individuals would give a precision of ± 5% to a point estimate equal to 15% of the prevalence of suicide risk at 30 days. Assuming a 10% refusal rate to participate in the follow-up visit, this number should be increased to 240 patients.

This number of 215 patients would give 80% power to a logistic regression model of the binary primary endpoint (Y, risk of suicide at 30 days) on a binary independent variable (X) in the presence of a binary covariate (Z). to detect, with an alpha risk of 0.05, an odds ratio equal to 2.50. This number is calculated under the assumption of a baseline risk for the primary endpoint Y of 0.15, the independence of observations, a prevalence of the independent variable X of 50%, a prevalence the covariate Z of 50% and an odds ratio of the primary endpoint Y associated with the covariate Z of 1.50. This number is calculated for a two-tailed Wald test.

The investigators believe that their study could have a real impact on CUMP practices and suicide risk prevention. In fact, the CUMP represents an original device and the context of the emergency and support groups may overlook the risk of suicide for some patients. In addition, there is currently no systematic monitoring planned within the CUMPs. It is therefore an innovative and particularly topical subject that could change clinical practices but also the organization of the healthcare offer. Indeed, several treatment centers for psychotrauma are currently being deployed at the national level (including a center in Lyon, within the Hospices Civils de Lyon (HCL)) and an important work of coordination of treatment structures is in progress.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for the first time by a CUMP directly confronted with a potentially traumatic event (PTE) (with ou without a previous psychiatric history)
* Patient affiliated with social welfare

Exclusion Criteria:

* Age under 18
* Not understanding French language.
* Not having provided the contact details of a trusted third party and of the attending physician
* Being homeless
* Information on the exhibition unavailable (subjects recently arrived in France, foreign language, etc.)
* A pathology requiring urgent medical treatment
* Covered by articles L1121-5 to L1121-8 of the CSP (pregnant women, parturients, breastfeeding women, persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric care and adults subject to a measure of legal protection or unable to express their consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients fulfilling the inclusion and non-inclusion criteria and having signed the consent will be included. Within 30 days (± 5 days), an appointment, by videoconference, will be made by the CUMP of the Grenoble center for the completion of the MINI scale and screening for suicidal behavior. This interview will be carried out either with the psychiatrist or the psychologist or with the psychiatric resident. If the patient does not answer, the trusted third party or the attending physician will be contacted by telephone in order to investigate the causes or to detect a possible death by suicide. The patient will be followed up one year after inclusion by telephone to detect the number of suicide attempts and/or death.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal risk | 30 days
  Absence or presence of the suicidal risk assessed using the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma

SECONDARY OUTCOMES:
Depressive disorders | 30 days
  Absence or presence of depressive disorders used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Bipolar disorders | 30 days
  Absence or presence of bipolar disorders used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Panic disorder | 30 days
  Absence or presence of panic disorders used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Agoraphobia | 30 days
  Absence or presence of agoraphobia used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Social phobia | 30 days
  Absence or presence of social phobia used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Generalized anxiety | 30 days
  Absence or presence of generalized anxiety used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Post-traumatic stress disorder | 30 days
  Absence or presence of post-traumatic stress disorder used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Obsessive-compulsive disorder | 30 days
  Absence or presence of obsessive-compulsive disorder used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Disorder linked to the consumption of alcohol or other substances | 30 days
  Absence or presence of disorder linked to the consumption of alcohol or other substances used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Psychotic disorders | 30 days
  Absence or presence of psychotic disorders used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Eating disorders | 30 days
  Absence or presence of eating disorders used the French transcultural adaptation of the Mini-International Neuropsychiatric Interview (MINI) after the possible psychological trauma
Mortality by suicide | 365 days
  Mortality by suicide after the psychological trauma (the cause of death is obtained from a trusted third party or from the attending physician)
Incidence of suicide | 365 days
  Number of patients having presented at least one suicide attempt during the 365 days after the psychological trauma (declaration of the patient or, in his absence, of the declared trusted person or the general practitioner)
Incidence of suicidal ideation | 365 days
  Number of patients declaring that they have presented suicidal ideation at least once during the 365 days after the psychological trauma (question yes / no)

CONTACTS AND LOCATIONS:
Overall Officials: Helene Poncet, MD, Principal Investigator — CHU Grenoble Alpes, SAMU38 - CUMP
Locations (4):
- France (4):
  - DELACHENAL Catherine, Chambéry
  - Geneste-Saelens, Clermont-Ferrand
  - VIGNAUD Philippe, Lyon
  - COURVOISIER Pierre, Montéléger